CLINICAL TRIAL: NCT03211117
Title: Phase 2 Study of Pembrolizumab Combined With Chemoradiation Therapy in Anaplastic Thyroid Cancer
Brief Title: Pembrolizumab, Chemotherapy, and Radiation Therapy With or Without Surgery in Treating Patients With Anaplastic Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1679; NCI-2017-01179 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1679 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-05

CONDITIONS: Thyroid Gland Undifferentiated (Anaplastic) Carcinoma
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — Docetaxel; Doxorubicin; Radiotherapy, Intensity-Modulated; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (pembrolizumab, surgery, chemoradiation) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients undergo surgery. Within 42 days of surgery, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Doxorubicin Hydrochloride; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Procedure: Therapeutic Conventional Surgery
- Cohort B (pembrolizumab, chemoradiation) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Doxorubicin Hydrochloride; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Cohort A (pembrolizumab, surgery, chemoradiation)

SUMMARY:
This phase II trial studies how well pembrolizumab, chemotherapy, and radiation therapy work with or without surgery in treating patients with anaplastic thyroid cancer. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as docetaxel and doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving pembrolizumab, chemotherapy, and radiation therapy with or without surgery may kill more tumor cells and work better in treating patients with anaplastic thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of pembrolizumab in improving overall survival at 6 months (OS-6) in combination with multimodal therapy involving standard chemo-radiotherapy in anaplastic thyroid cancer (ATC) in comparison to a historical cohort.

SECONDARY OBJECTIVES:

I. To determine safety and tolerance of pembrolizumab with chemoradiotherapy.

TERTIARY OBJECTIVES:

I. To evaluate locoregional control. II. To evaluate progression of distant metastases. III. To evaluate the evolution of the immune profile of circulating immune cells in response to therapy in ATC patents, and to assess potential correlations with outcomes on an exploratory basis.

IV. To evaluate PD-1 and PD-L1 staining in tumor cells and tumor stroma as candidate biomarkers for outcomes.

V. To determine if pre-therapy circulating tumor cell load is associated with outcomes.

VI. To examine associations between outcomes and somatic mutational status as assessed by foundation medicine analysis (for example: presence of BRAF, RAS, P53 and TERT promoter mutations).

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients undergo surgery. Within 42 days of surgery, patients also receive docetaxel IV over 1 hour once weekly (Q1W) and doxorubicin hydrochloride IV Q1W, and undergo intensity-modulated radiation therapy (IMRT) once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.

COHORT B: Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months until progressive disease and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of, or cytology reported and confirmed, anaplastic thyroid cancer

  * NOTE: A diagnosis reported as ?poorly differentiated carcinoma consistent with anaplastic thyroid cancer? will be accepted
* Absence of prior neck radiotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin >= 9.0 g/dL
* White blood cells (WBC)/leukocytes >= 3500/mm^3
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except for patients with well-documented Gilbert?s syndrome)
* Aspartate transaminase (AST) =< 3 x ULN
* Creatinine =< 1.5 x ULN OR calculated creatinine clearance >= 50 ml/min using the Cockcroft-Gault formula
* Prothrombin time (PT)/activated partial thromboplastin time (PTT) =< 1.5 x ULN, unless subject is receiving anticoagulant therapy and PT or activated (a)PTT is within therapeutic range of intended use of anticoagulants
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * NOTE: Merck requires an additional pregnancy test if eligibility pregnancy test is > 72 hours prior to first dose
* Persons of childbearing potential must be willing to use an adequate method of birth control for the course of the study through 120 days after the last dose of study medication

  * NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred method of contraception for the patient
* Persons able to father a child must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred method of contraception for the patient
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* History of non-infectious pneumonitis that required steroids or current pneumonitis
* Any of the following:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Any autoimmune disease such as inflammatory bowel disease, including but not limited to:

  * Ulcerative colitis
  * Crohn's disease
  * Rheumatoid arthritis
  * Systemic sclerosis
  * Systemic lupus erythematosus
  * Autoimmune hepatitis
  * Other autoimmune disease not listed above
  * NOTE: Subjects with autoimmune thyroid disease and diabetes mellitus type I will be allowed
* Uncontrolled intercurrent illness including, but not limited to,

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia, or
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Other active malignancy =< 6 months prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix or prostate cancer confined to prostate gland with Gleason score < 6 or prostate-specific antigen (PSA) < 1
  * NOTE: If there is a history of prior malignancy, they must not be receiving other treatment for their cancer; ongoing adjuvant hormonal treatment for breast cancer is allowed
* Prior known allergic reaction to pembrolizumab or its excipients
* Untreated brain metastasis
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Received any live vaccine =< 30 days prior to registration
* Any of the following conditions =< 6 weeks prior to registration:

  * Cerebrovascular accident (CVA)
  * Admission for unstable angina
  * Cardiac angioplasty or stenting or coronary artery bypass graft surgery
  * Pulmonary embolism or untreated deep venous thrombosis (DVT)
  * Arterial thrombosis
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Chintakuntlawar, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (Pembrolizumab, Surgery, Chemoradiation): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients undergo surgery. Within 42 days of surgery, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.
  Docetaxel: Given IV Doxorubicin Hydrochloride: Given IV Intensity-Modulated Radiation Therapy: Undergo IMRT Laboratory Biomarker Analysis: Correlative studies Pembrolizumab: Given IV Therapeutic Conventional Surgery: Undergo surgery
- Cohort B (Pembrolizumab, Chemoradiation): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.
  Docetaxel: Given IV Doxorubicin Hydrochloride: Given IV Intensity-Modulated Radiation Therapy: Undergo IMRT Laboratory Biomarker Analysis: Correlative studies Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Cohort A (Pembrolizumab, Surgery, Chemoradiation) | Cohort B (Pembrolizumab, Chemoradiation)
Started | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort B (Pembrolizumab, Chemoradiation): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.>
  > Docetaxel: Given IV>
  > Doxorubicin Hydrochloride: Given IV>
  > Intensity-Modulated Radiation Therapy: Undergo IMRT>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Pembrolizumab: Given IV
Arm/Group | Cohort B (Pembrolizumab, Chemoradiation)
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 56 [55 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate
Description: Defined as the percentage of evaluable patients who are alive at 6 months.
Time Frame: At 6 months
Population: All patients
Measure: Number; unit: percentage of participants alive
Arm/Group | Cohort B (Pembrolizumab, Chemoradiation)
Number analyzed (Participants) | 3
percentage of participants alive | 0

2. Secondary Outcome: Incidence of Adverse Events Graded Using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine adverse event patterns. This data is reported in the adverse events section of this report.
Time Frame: 2.3 years
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B (Pembrolizumab, Chemoradiation): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.
  >
  > Docetaxel: Given IV
  >
  > Doxorubicin Hydrochloride: Given IV
  >
  > Intensity-Modulated Radiation Therapy: Undergo IMRT
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Pembrolizumab: Given IV
Arm/Group | Cohort B (Pembrolizumab, Chemoradiation)
Number analyzed (Participants) | 3
Participants | 3

3. Other Pre Specified Outcome: Number of Patients With Locoregional Recurrence and Locoregional Progression in the Thyroid Bed or Regional Lymph Nodes
Description: Will be summarized using descriptive statistics.
Time Frame: 2.3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Pembrolizumab, Chemoradiation)
Number analyzed (Participants) | 3
Participants | 0

4. Other Pre Specified Outcome: Numbers of Patients With Distant Metastasis
Description: Will be summarized using descriptive statistics.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2.3 years
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Groups:
- Cohort A: Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 21 days for up to 17 courses after chemoradiation if no residual disease is found or for up to 35 courses after chemoradiation if residual disease is found. After 3 days, patients undergo surgery. Within 42 days of surgery, patients also receive docetaxel IV over 1 hour Q1W and doxorubicin hydrochloride IV Q1W, and undergo IMRT once daily 5 days per week for 6.5 weeks in the absence of disease progression or unacceptable toxicity.
  Docetaxel: Given IV Doxorubicin Hydrochloride: Given IV Intensity-Modulated Radiation Therapy: Undergo IMRT Laboratory Biomarker Analysis: Correlative studies Pembrolizumab: Given IV Therapeutic Conventional Surgery: Undergo surgery
Arm/Group | Cohort B (Pembrolizumab, Chemoradiation) | Cohort A
All-Cause Mortality (participants affected / at risk) | 3/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort B (Pembrolizumab, Chemoradiation) (N=3) | Cohort A (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort B (Pembrolizumab, Chemoradiation) (N=3) | Cohort A (N=0)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (7) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 2 (5) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03211117/Prot_SAP_000.pdf